CLINICAL TRIAL: NCT03193138
Title: Cardiotoxicity of Androgenic Agonists and Antagonists in the National French Pharmacovigilance Database and EudraCT Database
Brief Title: CardioTOxicity Induced by andRogeNICS and Their Antagonists (TORNICS)
Acronym: TORNICS
Status: Completed | Type: Observational
Sponsor: Groupe Hospitalier Pitie-Salpetriere (Other)
Responsible Party: Principal Investigator, Joe Elie Salem, MD, PhD, Groupe Hospitalier Pitie-Salpetriere
Other Study IDs: CIC1421-17-06
Record Dates: First submitted 2017-06-12; First posted 2017-06-20 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Heart Diseases
Keywords: Cardiotoxicity; Androgens; Hormone Replacement Therapy; Testosterone; Androgen Antagonists
MeSH Terms: conditions — Heart Diseases; Cardiotoxicity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Hormonal therapies: G03, H01C and L02 in the ATC classification — Hormonal therapies including all therapies classified G03, H01C and L02 in the ATC classification

SUMMARY:
Anti-androgenic therapies relying on peripheral and/or central blockade for the treatment of prostate cancer seems to have an impact on the cardio-vascular system. This study investigates reports of cardiovascular toxicities for treatment including Anatomical Therapeutic Chemical (ATC) classification: sex hormones (G03), hypothalamic hormones (H01C) and sex hormones used in treatment of neoplastic diseases (L02) in the French pharmacovigilance database and European Clinical Trials (EudraCT) database.

DETAILED DESCRIPTION:
Hormone replacement therapies and contraceptive pills are responsible of a wide range of cardio-vascular side effects, particularly thrombo-embolic disorders and ischemic heart disease. The difference of incidence and type of cardio-vascular events between men and women are strongly related to sex hormones. Androgenic agonists and antagonists are used in various indication including prostate cancer or hormone replacement therapies. This study investigates the main characteristics of patients affected by cardiovascular side effects (of which ventricular arrhythmia's, QT prolongation and Torsade de Pointe) imputed to drugs classified as G03, H01C and L02 according to ATC. A causality assessment according to both Begaud's method and the World Health Organization-The Uppsala Monitoring Centre (WHO-UMC) is systematically applied.

ELIGIBILITY:
Inclusion Criteria:

* Case reported in the French pharmacovigilance database and EudraCT database from 01/01/1985 to 14/04/2017
* Adverse event reported were including the MedDRA terms: SOC Cardiac Affections and the HLT Death and Sudden Death
* Patients treated with hormonal therapies included in the ATC classification references: G03, H01C and L02

Exclusion Criteria:

* Chronology not compatible between the drug and the toxicity

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male
Study Population: The population is selected in the French pharmacovigilance database and EudraCT database from 01/01/1985 to 14/04/2017 and included patients treated with hormonal therapies included in the ATC classification references: G03, H01C and L02.
Sampling Method: Non-Probability Sample
Enrollment: 3096 (Actual)
Dates: Start 2017-06-07 (Actual); Primary Completion 2017-06-21 (Actual); Study Completion 2017-06-21 (Actual)

PRIMARY OUTCOMES:
Identification and report of the cardio-vascular toxicity of anti-androgenic therapies (reference G03 in the ATC classification) with a causality assessment using Begaud's and WHO's method. | Immediate evaluation
  The research includes the report with MedDRA terms: System Organ Class (SOC) Cardiac Disorders and High Level Term (HLT) Death and Sudden Death. Drugs investigated are hormonal therapies with the reference G03 in the ATC classification
Identification and report of the cardio-vascular toxicity of anti-androgenic therapies (reference H01C in the ATC classification) with a causality assessment using Begaud's and WHO's method. | Immediate evaluation
  The research includes the report with MedDRA terms: System Organ Class (SOC) Cardiac Disorders and High Level Term (HLT) Death and Sudden Death. Drugs investigated are hormonal therapies with the reference H01C in the ATC classification
Identification and report of the cardio-vascular toxicity of anti-androgenic therapies (reference L02 in the ATC classification) with a causality assessment using Begaud's and WHO's method. | Immediate evaluation
  The research includes the report with MedDRA terms: System Organ Class (SOC) Cardiac Disorders and High Level Term (HLT) Death and Sudden Death. Drugs investigated are hormonal therapies with the reference L02 in the ATC classification

SECONDARY OUTCOMES:
Causality assessment of reported cardiovascular events | Immediate evaluation
  Causality assessment of reported cardiovascular events according to the WHO-UMC system
Type of cardiotoxicity depending on the category and type of hormonal therapy | Immediate evaluation
  Description of the type of cardiotoxicity depending on the category and type of hormonal therapy
Duration of treatment when the toxicity happens | Immediate evaluation
  Description of the duration of treatment when the toxicity happens (role of cumulative dose)
Drug-drug interactions associated with adverse events | Immediate evaluation
  Description of the drug-drug interactions associated with adverse events (particularly heart failure, ischemic heart disease and cardiac arrhythmia's)
Pathologies for which the incriminated drugs have been prescribed | Immediate evaluation
  Description of the pathologies (cancer, hormonal insufficiency) for which the incriminated drugs have been prescribed
Population of patients having a cardio-vascular adverse event | Immediate evaluation
  Description of the population of patients having a cardio-vascular adverse event

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Régional de Pharmaco-vigilance - Paris, Pitié-Salpétrière, Paris, Île-de-France Region, France

REFERENCES:
- [Background] Salem JE, Yang T, Moslehi JJ, Waintraub X, Gandjbakhch E, Bachelot A, Hidden-Lucet F, Hulot JS, Knollmann BC, Lebrun-Vignes B, Funck-Brentano C, Glazer AM, Roden DM. Androgenic Effects on Ventricular Repolarization: A Translational Study From the International Pharmacovigilance Database to iPSC-Cardiomyocytes. Circulation. 2019 Sep 24;140(13):1070-1080. doi: 10.1161/CIRCULATIONAHA.119.040162. Epub 2019 Aug 5. PMID 31378084
- [Result] Salem JE, Waintraub X, Courtillot C, Shaffer CM, Gandjbakhch E, Maupain C, Moslehi JJ, Badilini F, Haroche J, Gougis P, Fressart V, Glazer AM, Hidden-Lucet F, Touraine P, Lebrun-Vignes B, Roden DM, Bachelot A, Funck-Brentano C. Hypogonadism as a Reversible Cause of Torsades de Pointes in Men. Circulation. 2018 Jul 3;138(1):110-113. doi: 10.1161/CIRCULATIONAHA.118.034282. No abstract available. PMID 29967236
- [Result] Barber M, Nguyen LS, Wassermann J, Spano JP, Funck-Brentano C, Salem JE. Cardiac arrhythmia considerations of hormone cancer therapies. Cardiovasc Res. 2019 Apr 15;115(5):878-894. doi: 10.1093/cvr/cvz020. PMID 30698686
- [Derived] Salem JE, Yang T, Moslehi JJ, Waintraub X, Gandjbakhch E, Bachelot A, Hidden-Lucet F, Hulot JS, Knollmann BC, Lebrun-Vignes B, Funck-Brentano C, Glazer AM, Roden DM. Androgenic effects on ventricular repolarization: A translational study from the international pharmacovigilance database to iPSC-cardiomyocytes. Ann Endocrinol (Paris). 2021 Jun;82(3-4):132-133. doi: 10.1016/j.ando.2020.02.008. Epub 2020 Feb 29. PMID 32171470